CLINICAL TRIAL: NCT02410421
Title: Validation of Individualized rTMS Protocol Using Non Invasive Functional Brain Imaging and Robotic Coil Placement in Resistant Depression: Comparison With Classical rTMS and tDCS
Brief Title: e-PAT Neuromod Evaluation of Personalized rTMS for Resistant Depression
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5055
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Depressive Disorder; Treatment-Resistant
Keywords: Individualized Medicine; Functional Neuroimaging; Robotic Proceedure; Transcranial Magnetic Stimulation, Repetitive; Transcranial Direct Current Stimulation Monocentric; Compariative Cross-Over 3 Arms Study Randomized, Single-Blind Method
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Individualized rTMS protocol (Experimental): The target region will be defined by comparing the rCBF scan of the patient to a control population (n = 80). rCBF will be measured using the QUIPS2 arterial spin labeling sequence on a Siemens 3T Verio.
  The therapeutic protocol will be design to correct the rCBF anomaly first by defining each point where to deliver the stimulation than the stimulation protocol for each point (180% of active motor threshold, 4-second 10 Hz train duration, with 26-second intertrain interval for a total of 3000 pulses). The whole target will be homogeneously stimulated.
  The active motor threshold will be assessed. The programmed protocol will be delivered while a figure of eight coil will be positioned by a robotic device (Axilum Robotics).
  The procedure will be repeated twice a day for 10 days over 2 weeks.
  Interventions: Procedure: Functional magnetic resonance imaging used to individualize rTMS protocol using robotic coil positioning
- High frequency rTMS as usual (Active Comparator): rTMS will be performed as usual using a figure-eight coil: Defining the active motor threshold. For each session positioning the coil 5 cm ahead of the abductor pollicis brevis muscle, stimulating at 180% of active motor threshold (10 Hz, 4-second train duration, and 26-second intertrain interval) for 37.5 minutes (3000 pulses per session), twice a day for 10 days over 2 weeks.
  Coil and stimulator will remain the same between individualized and "as usual" proceedures.
  Interventions: Procedure: Functional magnetic resonance imaging used to individualize rTMS protocol using robotic coil positioning
- Trans-cranial direct current stimulation (tDCS) (Active Comparator): tDCS will be performed as usual: After controlling for skin healthiness, the anode and the cathode will be respectively placed over F3 and F4. A commercial devices (MagStim), will deliver a constant current of 2 mA through 25 cm2 saline-soaked rubber sponges for 20 min per session. The procedure will be repeated twice a day for 10 days over 2 weeks.
  Interventions: Procedure: Functional magnetic resonance imaging used to individualize rTMS protocol using robotic coil positioning

INTERVENTIONS:
Procedure: Functional magnetic resonance imaging used to individualize rTMS protocol using robotic coil positioning

SUMMARY:
Although repetitive trans-cranial magnetic stimulation (rTMS) is an effective therapy for resistant depression, it still fail to remit up to 70% of these patients. We hypothesize that personalizing the procedure using functional MRI to better select dysfunctional regions and robotic coil placement to stimulate these regions homogeneously, will increase its efficacy. Individualized rTMS will be compared to traditional rTMS procedure and to trans-cranial direct current stimulation (tDCS).

In this small proof of principle study our primary outcome measure will be the correction of the MRI anomalies. Symptoms reduction and the proportion of remitters will be secondary outcome measurements.

ELIGIBILITY:
Inclusion criteria:

* Aged from 18 to 65 Y
* Affiliated to the health insurance
* Having signed an informed consent
* Suffering from major depression according to the DSM5
* Unresponsive or incomplete remission after at least one trial of antidepressant (> 6 weeks at efficient dose or side effects)
* Treatment stable for > 6 weeks

Exclusion criteria:

* Contraindication for MRI, rTMS or tDCS: non-removable ferromagnetic body, prosthesis, pacemaker, medication delivered by an implanted pump clip or vascular stent, heart valve or ventricular shunt, seizure disorders, skin pathology in the region of tDCS electrode placement.
* Pregnancy
* Severe and non-stabilized somatic pathology
* Patients deprived of liberty or hospitalized without their consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Reduction of the target regional cerebral blood flow (rCBF) anomaly | difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  The target region will be defined by comparing the rCBF scan of the patient to a control population (n = 80). rCBF will be measured using the QUIPS2 arterial spin labeling sequence on a Siemens 3T Verio. We will compare the average rCBF of the target region before and after the therapeutic protocol between the different procedures (ANOVA).
Reduction of the functional connectivity anomalies | difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  Functional connectivity map of the target region will be performed by extracting its average temporal course and looking at the region(s) which activity is correlated (smoothed by a 8 mm Gaussian kernel). The contrast map of each patient will be compared to the one of a control population submitted to the same analysis. We will compare the number of above threshold voxels (F-test, p < 0.05 uncorrected, extension > 1 cm3) before and after the therapeutic procedure (ANOVA). We will compare the average rCBF of the target region before and after the therapeutic protocol between the different procedures (ANOVA).

SECONDARY OUTCOMES:
Symptoms evaluated by the clinician (QIDS16-C) | difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  See http://www.ids-qids.org/ for documentation relative to these scales.
  Computation will be performed in terms of :
  * Percentage of symptom reduction
  * Number responders (reduction of more than 50% of symptoms)
  * Numbers of remitters (QIDS16-C ≤ 6).
Symptoms evaluated by the patient (QIDS30-SR) | difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  See http://www.ids-qids.org/ for documentation relative to these scales.
  Computation will be performed in terms of :
  * Percentage of symptom reduction
  * Number responders (reduction of more than 50% of symptoms)
  * Numbers of remitters (QIDS16-C ≤ 6).

OTHER OUTCOMES:
Response time and accuracy at the attentional network test | Difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  * Switch or mixed states (MAThyS)
  * NAA/Choline and Lactate of the target (NMR spectroscopy)
Quality of life ("Echelle synoptique des 3 temps") | difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  * Switch or mixed states (MAThyS)
  * NAA/Choline and Lactate of the target (NMR spectroscopy)
Global Assessment of Functioning | Difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  * Switch or mixed states (MAThyS)
  * NAA/Choline and Lactate of the target (NMR spectroscopy)
Activity measured by an actimeter | Difference between before (D-7 to -1) and after (D+15 to +21) each therapeutic protocol (D = day of the beginning of the protocol)
  * Switch or mixed states (MAThyS)
  * NAA/Choline and Lactate of the target (NMR spectroscopy)
Acceptance of each therapeutic procedure | We will directly compare each therapeutic protocol by averaging this value from D1 to D12.
  Feeling comfortable with the environment (visual analog scale), this will be evaluated at each stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Jack FOUCHER, MD, Principal Investigator — Service de Psychiatrie 1, Hôpitaux Universitaires de Strasbourg